CLINICAL TRIAL: NCT06978829
Title: Cetuximab Combined With Tislelizumab and Chemotherapy in the Treatment of Unresectable Locally Advanced Head and Neck Squamous Cell Carcinoma: A Prospective, Single-Arm, Phase II Study
Brief Title: Cetuximab + Tislelizumab + Chemotherapy in the Treatment of Unresectable LA HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202552
Record Dates: First submitted 2025-04-16; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-02

CONDITIONS: LA HNSCC
Keywords: Tislelizumab; Cetuximab; LA HNSCC
MeSH Terms: interventions — Cetuximab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Conversion therapy stage：TP+Cetuximab+Tislelizumab. Radical therapy stage: Those assessed as operable receive curative surgery, while those assessed as inoperable undergo radical radiotherapy.
  Maintenance therapy stage: Tislelizumab for 1 year.
  Interventions: Drug: TP + Cetuximab + Tislelizumab

INTERVENTIONS:
Drug: TP + Cetuximab + Tislelizumab — Conversion therapy stage:
  TP regimen: Albumin-bound paclitaxel+Platinum (Cisplatin or Carboplatin) Albumin-bound paclitaxel: 100 mg/m² by IV infusion, D1/D8, every 3 weeks (Q3W) Platinum: Cisplatin 75 mg/m² by IV infusion or Carboplatin AUC=5 mg/mL/min Q3W Cetuximab: The initial dose is 400 mg/m² by IV infusion for 1 week. Subsequently followed by 250 mg/m² IV infusion, D1/D8, Q3W.
  Tislelizumab: 200 mg by IV infusion, Q3W. 3 weeks/cycle, 3 cycles in total.
  Patients who have completed conversion therapy undergo efficacy evaluation.
  Radical therapy stage:
  Evaluated as operable: Undergo surgery, followed by one cycle of adjuvant chemotherapy according to the preoperative regimen.
  Evaluated as inoperable: Receive radical radiotherapy.
  Maintenance therapy stage:
  Tislelizumab for 1 year or until disease progression, intolerable toxicity, or patient refusal to continue treatment.

SUMMARY:
This prospective, single-arm, Phase II study aims to evaluate the efficacy, safety, and surgical conversion rate of Cetuximab combined with Tislelizumab and chemotherapy for unresectable LA HNSCC.

DETAILED DESCRIPTION:
This study plans to enroll 42 patients. After screening and qualifying the patients, they will be given the treatment of Cetuximab combined with Tislelizumab and the TP chemotherapy regimen. One cycle lasts for 3 weeks, and a total of 3 cycles will be carried out, followed by efficacy evaluation.

1. Patients evaluated as resectable will undergo surgical treatment. After the surgery, based on the postoperative pathology, it will be determined whether radiotherapy is needed. And then, 1 cycle of combined chemotherapy will be continued, followed by 1 - year maintenance treatment with Tislelizumab.
2. Patients evaluated as unsuitable for surgery will receive radical radiotherapy, followed by 1 - year maintenance treatment with Tislelizumab, until disease progression, intolerable adverse reactions occur, or the patient refuses to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates, signs the Informed Consent Form (ICF), and is able to comply with the study procedures;
2. Patients with locally advanced head and neck squamous cell carcinoma confirmed by cytology or histology, for whom complete surgical resection is difficult;
3. No prior treatment for head and neck squamous cell carcinoma;
4. No prior treatment with cetuximab or PD-(L)1 inhibitors;
5. At least one measurable lesion according to RECIST v1.1;
6. No gender restriction, age ≥18;
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
8. Expected survival period ≥ 3 months;
9. Organ function levels meet the following criteria:

   1. Blood routine: Hemoglobin ≥90 g/L, absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥90×10^9/L;
   2. Blood biochemistry: ALT, AST ≤2.5×ULN (≤5×ULN if liver metastasis is present), total serum bilirubin ≤1.5×ULN, serum creatinine ≤1.5×ULN, serum albumin ≥30 g/L;
   3. Cardiac function: Left ventricular ejection fraction >50% as shown by echocardiography.
10. Women of childbearing potential must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and be willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the trial drug.

Exclusion Criteria:

1. Previous anti-tumor treatments received (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Known or suspected allergy to any component of cetuximab or PD-(L)1 monoclonal antibodies, as well as to the chemotherapeutic drugs paclitaxel and cisplatin;
3. Patients with hypertension that cannot be controlled to normal range with antihypertensive medications (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg), patients with coronary heart disease of grade II or above, grade II arrhythmia (including QTc interval prolongation >470 ms), and grade I cardiac insufficiency;
4. History of autoimmune diseases or autoimmune disease history (such as colitis, hepatitis, hyperthyroidism, including but not limited to these diseases or syndromes), immunodeficiency history, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation;
5. Uncontrolled active hepatitis B (HBV DNA ≥ 1000 IU/mL) or active hepatitis C (positive hepatitis C antibody) patients;
6. Patients with active tuberculosis (with exposure history or positive tuberculosis test; accompanied by clinical and/or imaging manifestations);
7. Patients who have undergone major surgery within 4 weeks before the first dose or whose wounds have not fully healed;
8. Patients with a clear tendency to bleed;
9. Patients with severe complications such as pyloric obstruction, upper gastrointestinal bleeding, gastrointestinal perforation, obstructive jaundice, severe malnutrition, etc.;
10. Patients who have experienced abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months before enrollment;
11. Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the patient's tumor is highly likely to invade important blood vessels during treatment, leading to fatal massive bleeding;
12. History of interstitial lung disease, non-infectious pneumonia, or uncontrolled diseases, including pulmonary fibrosis, acute lung disease, etc.;
13. Patients with active brain metastasis;
14. Patients with other malignant tumors within 5 years (except for completely cured cervical carcinoma in situ or basal cell or squamous cell skin cancer);
15. Pregnant or breastfeeding women;
16. Patients with severe concomitant diseases that endanger patient safety or affect the completion of the study, as judged by the investigator, and those whom the investigator considers unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  Defined as the proportion of participants acquired Complete response (CR) or Partial response (PR) after conversion treatment. Based on RECIST 1.1.

SECONDARY OUTCOMES:
R0 resection rate | 6 months
  Defined as the proportion of patients in whom no cancer cells are detected at the resection margin microscopically, with no residual cancer cells visible either macroscopically or microscopically, and the lesion is completely excised.
Major Pathological Response Rate (MPR) | 6 months
  Defined as the presence of 10% or less viable tumor cells in the resected specimen following preoperative therapy, as assessed by pathological examination.
Progression free survival (PFS) | up to 5 years
  Defined as the period from enrollment to disease progress or death.
Overall Survival (OS) | up to 5 years
  Defined as the period from enrollment to death from any cause
Adverse Event rate | up to 2 years
  The rate of adverse event after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided